CLINICAL TRIAL: NCT05483686
Title: Reducing HIV Health Disparities Among African American Transgender Women: An mHealth Approach to Improving Prevention, Testing, and Treatment Outcomes
Brief Title: Improving HIV Outcomes Among African American Transgender Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ISA Associates, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R44MH117837 (NIH)
Record Dates: First submitted 2022-07-15; First posted 2022-08-02 (Actual); Results first posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: HIV
MeSH Terms: interventions — quadrant anterior shine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shine Intervention (Experimental): Experimental group participants will have access to the mobile Shine intervention.
  Interventions: Behavioral: Shine
- Control Videos (Active Comparator): Control condition participants will be texted an embedded link to a series of videos developed by the Centers for Disease Control. These videos describe healthy HIV-related behaviors for trans women of any status (e.g., recommended testing frequencies, PrEP, ART, condoms), includes videos of trans women describing their experiences with HIV. All control participants will have access to Shine at the end of the research study (i.e., approximately six months after recruitment).
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Shine — This tailored, multifaceted mobile intervention aims to improve HIV-related outcomes and increase gender affirmation among African American transgender women. Potential users will opt-in by texting from their own mobile phone and, once registered, will be enrolled into a program that will be theory-based, targeted, tailored, and personalized. Users will receive three main types of texts: informational, motivational, and skill-building. Finally, the program will include three web-based video components: scripted vignettes, unscripted peer narratives, and educational instruction. By developing an intervention using a technology that is part of the everyday lives of most African Americans, the aim is to reduce HIV disparities. The proposed intervention can be used by clinics and community-based organizations that serve transgender women.
  Arms: Shine Intervention
Behavioral: Control — A playlist of CDC-developed videos designed to provide information on HIV for transgender women
  Arms: Control Videos

SUMMARY:
The investigators will conduct a randomized controlled trial to test the efficacy of the mobile HIV behavioral intervention for African American transgender women (Shine). Participants will be 215 trans women recruited by staff of the Trans Women of Color Collective via community events and social media. Participants must : 1) identify as a Black transgender woman using the 2-step method (Step 1: assigned male birth sex, Step 2: current gender identity is female); 2) be aged 18 or older; 3) report risk of HIV transmission in past 3 months (i.e., CAS with a serodiscordant or risky partner AND either <90% ART adherence or <5 daily doses of PrEP per week); 4) own a smartphone; and 5) be able to read and speak English. Eligible participants who subsequently provide informed consent will complete two confidential phone-based research surveys at different time points (baseline and 6 months post-baseline) and will be randomly assigned to one of two conditions (Shine or mobile HIV education for transgender women).

Participants randomly assigned to the experimental condition will be instructed to text the word "Join" to the Shine study phone number. The intervention will take approximately 1-2 hours, with content delivered over several weeks. Participants randomly assigned to the control condition will be texted a link to a set of videos on healthy HIV-related behaviors for transgender women. These videos cover a variety of topics, including recommended testing frequencies, PrEP, and ART.

After randomization, participants will complete the baseline research survey. This survey will assess the primary outcome of composite HIV transmission risk along with several secondary outcomes (individual behavioral components of the composite score; HIV medical care utilization and adherence; HIV testing; PrEP knowledge, interest, and uptake; gender affirmation; well-being; social support; sexual communication). Six months after the baseline research survey, all participants will complete a follow-up research survey assessing the same outcome measures in the baseline research survey.

Binomial logistic regression will be the main analytic technique for the primary measure (composite risk for HIV transmission). For the secondary continuous measures, hierarchical linear modeling (HLM) will be used. All models will control for any demographic covariate (e.g., age) that varies at the .2 significance level due to randomization failure at baseline.

DETAILED DESCRIPTION:
The investigators will conduct a randomized controlled trial to test the efficacy of Shine, an mHealth HIV behavioral intervention for African American transgender women (TGW). Participants will be 215 African American TGW recruited by Trans Women of Color Collective (TWOCC) via in-person and online recruitment strategies. First, TWOCC's leadership and administrative teams will distribute palm cards and display posters describing the study during all community-based events that occur during the recruitment period. Second, ISA and TWOCC will develop an online strategy to disseminate a study flyer via social media (e.g., Facebook, Twitter). The flyer will be posted on both social media channels weekly during the study recruitment period. Interested women recruited via either method (in-person or online) will be instructed to contact the ISA field test manager for more information and to complete eligibility screening.

Interested participants who contact the field test manager will complete an eligibility screener. Specifically, participants must : 1) identify as a Black transgender woman using the recommended 2-step method (Step 1: assigned male birth sex, Step 2: current gender identity is female); 2) be aged 18 or older; 3) report risk of HIV transmission in the past 3 months (i.e., CAS with a serodiscordant or risky male partner AND either <90% ART adherence or <5 daily doses of PrEP per week); 4) own a smartphone; and 5) be able to read and speak English.

Ineligible women will be thanked, dismissed, and offered alternatives to the type of information being offered in this research study. Eligible women will provide contact information receive a detailed overview of the main points of the study. Once any participant questions are answered, the field test manager will trigger a text to be sent to the potential participant's study phone number. The text will include a link to an online version of the informed consent form presented on a secure web page (i.e., communication between the phone's browser and web page are encrypted). Women who agree to participate will acknowledge consent by clicking a button at the bottom of the online consent form that reads "I understand and CONSENT to participate." Women who choose not to participate after reading the informed consent form will press a button that reads "I understand and choose NOT to participate." These women will be thanked and all contact will cease.

Participants will be assigned to conditions using a permuted-blocks randomization scheme. Blocks of size 4 and 6 will be used. Assignments within blocks will be random but balanced among the two conditions and the order of the blocks (4 vs 6) also will be random. This procedure will ensure that the number of participants randomized to each condition will be equal, that any imbalance among the conditions at any point during the recruitment and randomization will be modest, and that it will be very difficult to guess the assignment of the next participant. After randomization has occurred, participants will complete the baseline research survey via telephone.

The primary outcome will be a dichotomous composite HIV risk transmission score, calculated by measuring whether a participant or the participant's partner consistently used at least one effective method for reducing HIV transmission risk (i.e., adherence to biomedical [ART or PrEP] and behavioral [condoms, serosorting] strategies) during each instance of anal sex over the past month. Every anal sex act must be protected by one of these methods to receive an overall composite score of 0. The individual behavioral components of the composite score (i.e., percentage of condomless anal sex, serosorting, PrEP or ART adherence) will serve as secondary measures. In addition, specific outcomes by HIV status will include HIV medical care utilization and adherence, HIV testing, and PrEP knowledge, interest, and uptake. Finally, further secondary measures will assess gender affirmation, well-being, social support, and sexual communication.

Once the baseline research survey has been completed, participants will receive instructions for accessing the assigned materials. Those in the experimental group will be instructed to text the word "join" to the Shine study phone number. After joining, experimental group participants will be enrolled in a mobile intervention that aims to reduce HIV health disparities among African American TGW along the entire care continuum. Participants randomly assigned to the control condition will be texted a link to a set of videos on healthy HIV-related behaviors for transgender women. These videos cover a variety of topics, including recommended testing frequencies, PrEP, and ART. All control participants will have access to Shine at the end of the research study (i.e., approximately six months after recruitment).

Six months after the baseline research survey, all participants will complete a follow-up research survey assessing the same outcome measures in the baseline research survey.

Given a sample size of 215 and a predicted retention rate of 80%, the investigators anticipate having complete data for at least 172 participants at the close of the study. Because randomization carries the expectation of creating treatment groups equivalent with respect to known and unknown prognostic factors, removing randomized participants from the analysis runs the risk of tampering with this balance and introducing bias into the treatment comparisons. As a result, an intention-to-treat analytic approach will be followed such that all participants randomized into the study will be included in all analyses irrespective of protocol violations post randomization. Multiple imputation is now widely regarded as an effective method for replacing missing data, and the investigators will use this approach.

Binomial logistic regression will be the main analytic technique for the primary outcome (composite HIV transmission risk score) and other non-continuous measures. For continuous measures, hierarchical linear modeling (HLM) will be used. All models will control for any demographic covariate (e.g., age) that varies at the .2 significance level due to randomization failure at baseline.

To ensure this study will be fully powered, the investigators estimated power for the binomial logistic regression analysis on the binary primary outcome measure (composite HIV transmission risk score). To conduct this calculation, the investigators examined power from Garofalo and colleagues' RCT of LifeSkills, a 6-session group-based, in person intervention for young trans women of any HIV status. At the 12-month follow-up, TGW in the empowerment-based HIV intervention showed a 39.8% greater reduction in condomless sex compared to participants in a standard care control condition (risk ratio = .60). This effect is described as "robust" by the authors but is typically interpreted as a small-medium effect size (Cohen's d=.35). This study provides an adequate power comparison for two reasons. First, this intervention (empowerment-based) and population (specifically tailored for TGW) closely align with the proposed work. Second, this effect size is consistent with the average effect size of SMS-based interventions on health behaviors (d = .33). As the effect size for the binomial logistic regression is an odds ratio, the investigators translated the Cohen's d of .35 to an odds ratio of 1.89. The G*Power 3.1 program was then used to determine that an odds ratio of 1.89 and an α error probability of 0.05 requires a sample size of 172 to be sufficiently powered at 1-β error probability = 0.95. Therefore, the 172 participants the investigators expect to retain through the follow-up, given a sample size of 215 and a 20% attrition rate, should be sufficient to detect significant differences in composite risk for HIV transmission at follow-up.

ELIGIBILITY:
Inclusion Criteria:

* African American/Black
* identifies as a transgender woman using the recommended 2-step method (Step 1: assigned male birth sex, Step 2: current gender identity is female)
* 18 or older
* report risk of HIV transmission in past 3 months (i.e., CAS with a serodiscordant or risky partner AND either <90% ART adherence or <5 daily doses of PrEP per week)
* owns a mobile phone capable of SMS messaging and accessing webpages
* able to speak/understand English

Exclusion Criteria:

* does not meet inclusion criteria

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants must identify as a Black transgender woman using the recommended 2-step method (Step 1: assigned male birth sex, Step 2: current gender identity is female)
Enrollment: 38 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Leaf, Ph.D., Principal Investigator — ISA Associates
Locations (1):
- ISA Associates, Inc., Alexandria, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
The mode of dissemination of public datasets will be via archive files accessible in the public domain. Public datasets will be de-identified so that data cannot be linked to individual research participants.
Supporting Information: Study Protocol, SAP
Time Frame: Datasets will be available at a minimum once the data have been accepted for peer-reviewed publication, and earlier if the data are deemed by the PI to be clean and the sharing of data is not expected to inhibit future opportunities for publication.
Access Criteria: A data sharing agreement must be completed and signed by the requesting investigator and the Principal Investigator before this transfer of data can be made.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data were collected from 11/16/2021 - 1/30/2023 via telephone with participants recruited through online advertising
Pre-assignment Details: Of the 83 potential participants assessed for eligibility, 33 did not meet eligibility criteria and 12 did not return our calls to complete informed consent and enroll in the study.
Groups:
- Shine Intervention: Experimental group participants will have access to the mobile Shine intervention.
  Shine: This tailored, multifaceted mobile intervention aims to improve HIV-related outcomes and increase gender affirmation among African American transgender women. Potential users will opt-in by texting from their own mobile phone and, once registered, will be enrolled into a program that will be theory-based, targeted, tailored, and personalized. Users will receive three main types of texts: informational, motivational, and skill-building. Finally, the program will include three web-based video components: scripted vignettes, unscripted peer narratives, and educational instruction. By developing an intervention using a technology that is part of the everyday lives of most African Americans, the aim is to reduce HIV disparities. We envision the proposed intervention being used by clinics and community-based organizations that serve transgender women.
Period: Overall Study
Arm/Group | Shine Intervention | Control Videos
Started | 18 | 20
Completed | 13 | 13
Not Completed | 5 | 7
Not completed — Lost to Follow-up | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Shine Intervention | Control Videos | Total
Number analyzed (Participants) | 18 | 20 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.17 (9.20) | 35.90 (10.13) | 37.45 (9.71)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Transgender Woman | 18 | 20 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 20 | 38
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 20 | 38

OUTCOME MEASURES:

1. Primary Outcome: Change in Percentage of Participants With HIV Transmission Risk at Month 6
Description: Percentage of participants with a composite risk for HIV score of 1. The composite risk for HIV score combines participants' use of and adherence to biomedical and behavioral strategies over the past month into a binary indicator (0, 1) of HIV acquisition or transmission risk. 0 indicates some HIV transmission risk and 1 indicates no HIV transmission risk.
Time Frame: Baseline and Month 6
Measure: Number; unit: percentage of participants with no risk
Arm/Group | Shine Intervention | Control Videos
Number analyzed (Participants) | 13 | 13
percentage of participants with no risk
  Baseline | 23.077 | 38.462
  Month 6 | 46.154 | 46.154
Statistical Analysis 1: Comparison: Shine Intervention vs Control Videos; This analysis aims to detect a significant change (p = .05) in percentage of participants with HIV transmission risk between Shine Intervention participants and Control Videos participants from Baseline to Month 6; Test type: Superiority; p = .19, Regression, Logistic

2. Secondary Outcome: Change in ART Adherence at Month 6
Description: ART adherence was measured using the 8-item Morisky Medication Adherence Scale (MMAS-8). Total scores range from 0 ot 8 with higher scores indicating better adherence.
Time Frame: Baseline and Month 6
Population: Subsample of participants who completed the ART adherence measure (i.e., those who reported being currently prescribed ART).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Shine Intervention | Control Videos
Number analyzed (Participants) | 6 | 5
score on a scale
  Baseline | 3.38 (2.17) | 5.25 (1.26)
  Month 6 | 6.50 (1.29) | 6.50 (1.45)
Statistical Analysis 1: Comparison: Shine Intervention vs Control Videos; This analysis aims to detect a significant change (p = .05) in ART adherence between Shine Intervention participants and Control Videos participants from Baseline to Month 6; Test type: Superiority; p = .24, Mixed Models Analysis

3. Secondary Outcome: Change in Condom Use at Month 6
Description: Percentage of anal sex acts in the past month during which a condom was used
Time Frame: Baseline and Month 6
Measure: Mean (Standard Deviation); unit: percentage of sex acts with condom
Arm/Group | Shine Intervention | Control Videos
Number analyzed (Participants) | 13 | 13
percentage of sex acts with condom
  Baseline | 51.79 (36.68) | 49.39 (40.54)
  Month 6 | 37.33 (50.40) | 58.84 (41.74)
Statistical Analysis 1: Comparison: Shine Intervention vs Control Videos; This analysis aims to detect a significant change (p = .05) in condom use between Shine Intervention participants and Control Videos participants from Baseline to Month 6; Test type: Superiority; p = .79, Mixed Models Analysis

4. Secondary Outcome: Change in Barriers to ART Use at Month 6
Description: ART Barriers were measured with a 14-item measure developed by the Adult AIDS Clinical Trials Group; items rated on 0-4 Likert-type scale where higher scores indicate more barriers to ART use; min=0 and max=4 (averaged)
Time Frame: Baseline and Month 6
Population: Subsample of participants who completed the ART barriers measure (i.e., those who reported being currently prescribed ART).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Shine Intervention | Control Videos
Number analyzed (Participants) | 6 | 5
units on a scale
  Baseline | 1.02 (.79) | 1.04 (.41)
  Month 6 | .70 (.51) | .86 (.68)
Statistical Analysis 1: Comparison: Shine Intervention vs Control Videos; This analysis aims to detect a significant change (p = .05) in barriers to ART use between Shine Intervention participants and Control Videos participants from Baseline to Month 6; Test type: Superiority; p = .81, Mixed Models Analysis

5. Secondary Outcome: Change in Barriers to PrEP Use at Month 6
Description: 12 item scale (multiple choice) for HIV-negative or unknown status participants; items rated on 0-4 Likert-type scale where higher scores indicate more barriers to PrEP use; min=0 and max=4 (averaged)
Time Frame: Baseline and Month 6
Population: Subsample of participants who completed the PrEP barriers measure (i.e., those who reported being HIV-negative or of unknown HIV status).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Shine Intervention | Control Videos
Number analyzed (Participants) | 6 | 7
score on a scale
  Baseline | 2.62 (1.07) | 2.02 (1.39)
  Month 6 | 2.18 (.97) | 2.13 (1.47)
Statistical Analysis 1: Comparison: Shine Intervention vs Control Videos; This analysis aims to detect a significant change (p = .05) in barriers to PrEP use between Shine Intervention participants and Control Videos participants from Baseline to Month 6; Test type: Superiority; p = .14, Mixed Models Analysis

6. Secondary Outcome: Change in Barriers to Condom Use at Month 6
Description: 29-item scale (multiple choice); items rated on 0-4 Likert-type scale where higher scores indicate more barriers to condom use; min=0 and max=4 (averaged)
Time Frame: Baseline and Month 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Shine Intervention | Control Videos
Number analyzed (Participants) | 12 | 13
units on a scale
  Baseline | 1.20 (.68) | 1.09 (.97)
  Month 6 | 1.05 (.94) | .76 (.79)
Statistical Analysis 1: Comparison: Shine Intervention vs Control Videos; This analysis aims to detect a significant change (p = .05) in barriers to condom use between Shine Intervention participants and Control Videos participants from Baseline to Month 6; Test type: Superiority; p = .81, Mixed Models Analysis

7. Secondary Outcome: Change in Social Support at Month 6
Description: the 19-item Social Support Scale from the Medical Outcomes Study (multiple choice); items rated on 0-4 Likert-type scale where higher scores indicate greater social support; min=0 and max=4 (averaged)
Time Frame: Baseline and Month 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Shine Intervention | Control Videos
Number analyzed (Participants) | 13 | 13
units on a scale
  Baseline | 2.57 (1.06) | 2.68 (1.09)
  Month 6 | 2.86 (.94) | 2.53 (1.39)
Statistical Analysis 1: Comparison: Shine Intervention vs Control Videos; This analysis aims to detect a significant change (p = .05) in social support between Shine Intervention participants and Control Videos participants from Baseline to Month 6; Test type: Superiority; p = .30, Mixed Models Analysis

8. Secondary Outcome: Change in Gender Identity Comfort at Month 6
Description: measured using the 12-item Transgender Congruence Scale; 12 item scale (multiple choice); items rated on 0-4 Likert-type scale where higher scores indicate greater gender identity comfort; min=0 and max=4 (averaged)
Time Frame: Baseline and Month 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Shine Intervention | Control Videos
Number analyzed (Participants) | 13 | 13
units on a scale
  Baseline | 3.13 (.72) | 3.12 (.79)
  Month 6 | 3.17 (.70) | 3.13 (1.09)
Statistical Analysis 1: Comparison: Shine Intervention vs Control Videos; This analysis aims to detect a significant change (p = .05) in gender identity comfort between Shine Intervention participants and Control Videos participants from Baseline to Month 6; Test type: Superiority; p = .94, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 6 months (i.e., from the baseline assessment through the 6 month follow-up assessment)
Arm/Group | Shine Intervention | Control Videos
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/20
Other Adverse Events (participants affected / at risk) | 0/18 | 0/20

LIMITATIONS AND CAVEATS:
The number of participants recruited to the study was lower than the target sample size. Therefore, the analysis of the primary and secondary outcome measures were underpowered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/86/NCT05483686/Prot_SAP_000.pdf